CLINICAL TRIAL: NCT00759941
Title: A Comparison of Brinzolamide Ophthalmic Suspension, 1% (Azopt) TID vs. Placebo TID Added to Latanoprost Ophthalmic Solution, 0.005% (Xalatan) in Patients With Elevated IOP on a Prostaglandin
Brief Title: A Comparison of Azopt Versus Placebo Added to Xalatan in Patients With Elevated Intraocular Pressure (IOP) on a Prostaglandin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMA-07-08
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2012-07

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — brinzolamide; Ophthalmic Solutions; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xalatan + Azopt (Experimental): Xalatan dosed once a day at 10 pm, with Azopt dosed three times a day at 8 AM, 2 PM, and 10:05 PM as an adjunctive therapy for 3 months.
  Interventions: Drug: Brinzolamide 1% ophthalmic solution (Azopt); Drug: Latanoprost 0.005% ophthalmic solution (Xalatan)
- Xalatan + Placebo (Active Comparator): Xalatan dosed once a day at 10 pm, with placebo dosed three times a day at 8 AM, 2 PM, and 10:05 PM concomitantly for 3 months.
  Interventions: Drug: Placebo eye drops; Drug: Latanoprost 0.005% ophthalmic solution (Xalatan)

INTERVENTIONS:
Drug: Brinzolamide 1% ophthalmic solution (Azopt) — One drop three times a day in both eyes for 3 months
  Other Names: AZOPT
  Arms: Xalatan + Azopt
Drug: Placebo eye drops — One drop three times a day in both eyes for 3 months
  Arms: Xalatan + Placebo
Drug: Latanoprost 0.005% ophthalmic solution (Xalatan) — One drop once a day in both eyes for 3 months
  Other Names: Xalatan

SUMMARY:
The purpose of this study was to assess the efficacy of adding Azopt dosed three times a day to Xalatan as compared to that of adding placebo to Xalatan in patients with elevated intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral primary open angle glaucoma, ocular hypertension or pseudoexfoliation syndrome.
* Intraocular pressure greater than 18 mmHg (mean diurnal) and less than 32 mmHg.
* Other protocol-defined inclusion criteria applied.

Exclusion:

* Previous intraocular surgery, except uncomplicated clear cornea phacoemulsification or argon laser trabeculoplasty.
* Argon laser trabeculoplasty or phacoemulsification within the last 3 months.
* Central corneal thickness outside the 500 - 600 (inclusive) micron range as measured by ultrasonic pachymetry.
* Ocular or periocular inflammation within 3 months prior to study (except blepharitis related or seasonal allergic conjunctivitis).
* History of uveitis or previous intraocular inflammation (other than post-operatively).
* Hypersensitivity to sulfa, or benzalkonium chloride.
* History of use of any steroids for over 1 week within 3 months of screening or likely need for any corticosteroids during the study (except inhaled, nasal or topical non-ocular).
* Other protocol-defined exclusion criteria applied.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible glaucoma patients were recruited and enrolled from 7 US study sites between Oct 15, 2007 and April 06, 2009.
Pre-assignment Details: This reporting group includes all enrolled subjects.
Period: Overall Study
Arm/Group | Xalatan + Azopt | Xalatan + Placebo
Started | 42 | 44
Completed | 39 | 43
Not Completed | 3 | 1
Not completed — Use of medication | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Exited in error by site | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xalatan + Azopt | Xalatan + Placebo | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.90 (11.43) | 68.13 (11.59) | 65.58 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 15 | 19 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Intraocular Pressure, 8 AM, at 3 Months
Description: Intraocular pressure was measured by Goldmann applanation tonometry. A negative number indicated a reduction in intraocular pressure.
Time Frame: Day 0, 3 months
Population: All enrolled. Two subjects were excluded from the efficacy analysis due to an adverse event (1) and use of medication not permitted (1).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Xalatan + Azopt | Xalatan + Placebo
Number analyzed (Participants) | 40 | 44
mmHg | -3.13 (3.03) | -2.57 (2.63)

2. Primary Outcome: Mean Change From Baseline in Intraocular Pressure, 12 PM, at 3 Months
Description: as for outcome 1
Time Frame: Day 0, 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Xalatan + Azopt | Xalatan + Placebo
Number analyzed (Participants) | 40 | 44
mmHg | -3.30 (2.36) | -2.48 (2.92)

3. Primary Outcome: Mean Change From Baseline in Intraocular Pressure, 4 PM, at 3 Months
Description: as for outcome 1
Time Frame: Day 0, 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Xalatan + Azopt | Xalatan + Placebo
Number analyzed (Participants) | 40 | 44
mmHg | -3.00 (3.40) | -2.33 (3.18)

4. Primary Outcome: Mean Change From Baseline in Intraocular Pressure, Diurnal, at 3 Months
Description: Diurnal intraocular pressure is the mean of the three timepoints measured (8AM, 12PM & 4PM). Intraocular pressure was measured by Goldmann applanation tonometry. A negative number indicated a reduction in mean intraocular pressure.
Time Frame: Day 0, 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Xalatan + Azopt | Xalatan + Placebo
Number analyzed (Participants) | 40 | 44
mmHg | -3.20 (2.55) | -2.48 (2.37)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 15-OCT-2007 to 31-JUL-2009.
Description: The safety population included all enrolled and exposed subjects.
Arm/Group | Xalatan + Azopt | Xalatan + Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/44
Other Adverse Events (participants affected / at risk) | 0/42 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.